CLINICAL TRIAL: NCT04224168
Title: Pectin Use in Pediatric Intestinal Rehabilitation: Comparison Study of Liquid Pectin Versus Green Beans in Optimizing Enteral Nutrition in Short Bowel Syndrome Patients
Brief Title: Pectin Use in Pediatric Intestinal Rehabilitation
Acronym: PUPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Le Bonheur Children's Hospital (Other)
Collaborators: University of Tennessee (Other)
Responsible Party: Principal Investigator, Meredith L Harvie, MD, Principal Investigator, Le Bonheur Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-06654-FB
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green Beans (Experimental): Green beans will be provided in the daily diets of the patients enrolled for 3 months via gtube or oral means. Only up to 6g of fiber total from green beans will be given. This equates to 3x 4 ounce jars of green beans per day.
  Interventions: Dietary Supplement: Green Beans
- Liquid Pectin (Experimental): Liquid pectin will be provided in the daily diets of the patients enrolled for 3 months via gtube or oral means. Only up to 6g of fiber total from liquid pectin will be given. This equates to 6 teaspoons or 30mL of liquid pectin per day.
  Interventions: Dietary Supplement: Liquid Pectin

INTERVENTIONS:
Dietary Supplement: Green Beans — Please see arm group Green beans for description
  Arms: Green Beans
Dietary Supplement: Liquid Pectin — Please see arm group liquid pectin for description
  Arms: Liquid Pectin

SUMMARY:
Pediatric short bowel patients, age 6 months to 21 years old, followed in our intestinal rehabilitation clinic, will be screened for qualification in the study. If meets qualification, will be consented for the study. The study involves patients receiving green beans in their diet for three months with data collection including stooling patterns as well as labs, and then switching over to liquid pectin for three months. Again data collection will take place. The duration of the study once patient is consented is ~6 months.

DETAILED DESCRIPTION:
This will be a modified cross over design. Patients who meet eligibility criteria, will be consented in their standard of care intestinal rehab clinic visit. Due to the fact that some patients who qualify for the study may already be on liquid pectin prior to the study, we will not be able to randomize all of the patients prior to starting the intervention. If a patient is on liquid pectin, they will stay on liquid pectin as their first intervention. If the patient is on no form of daily pectin, they will be randomized to either green beans or liquid pectin first. The patient will either be given Ball real fruit liquid pectin, 1g fiber/tsp, (mixed in formula or other liquid) via oral route or gastric tube (gtube) or Gerber stage two green bean baby food, 2gfiber/jar, via oral route or gtube. We will have patients stay on either Ball real fruit liquid pectin or Gerber stage 2 green beans for three months. After the three-month trial on one of the pectin formulation, they will switch to the other. However, we will not start collecting data until a week after the switch to allow for a washout period without compromising potential benefit that the patient was receiving. Each patient will receive 2g/kg of fiber per day(based on previous case reports) with a max of 6g/day. Patients will be followed in the Children's Intestinal Rehabilitation Clinic at Le Bonheur (CIRCLe). Standard of care follow up for short bowel syndrome patients is three months if they are doing well. During the three months, families will be contacted every 4 weeks via patient portal or phone call to ask specific questions on their current form of pectin, amount, days missed, ease/difficulty of administration and clinical symptoms. This will also serve as a reminder to the parents of what they should be providing to the child and will assist in optimizing data collection. After three months of being on one formulation of pectin, they will change to the other formulation and same follow up will occur. Stool output data collection will be delayed one week in between interventions as detailed above to allow for a "wash out" period. Standard of care also includes lab work (complete metabolic panel, magnesium, phosphorous, triglyceride, complete blood count with differential) at each 3 month visit. Trace minerals and soluble vitamins are usually collected annually, but for this study, will plan to obtain serum copper and iron levels after each intervention(x2). However, additional venous puncture will not be required. Therefore, data can be collected prior to intervention and following each intervention, then be compared between the groups. If able, we will collect stool samples from patients prior to intervention and after intervention to evaluate the microbiome. Recruitment in the study would be for a total period of six months. Interventions would be completed over a six month period. This allows us a total of 12 months for recruitment, intervention and data collection.

ELIGIBILITY:
Inclusion criteria:

* Short bowel syndrome patients followed in CIRCLe
* >=50% of colon remaining
* Patients requiring only enteral feeds for nutrition
* >=6 months of age-21 years of age

Exclusion criteria:

* Patients with major structural cardiac anomalies and/or end stage renal disease
* Patients with solid organ transplant
* Patients >24 months of age without gastric tube
* Short bowel patients on PN

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Weight gain | 6 months
  Z-score will be used to evaluate overall weight gain. This will standardize weight between ages. Weight will be taken prior to intervention and after each intervention.
Stooling pattern | 6 months
  Will use postcards to characterize stooling consistency and amount of stool. They will be weekly postcards that are mailed back to the clinic. Will take the average consistency and amount each week and compare before and after each intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anushree Algotar, MBBS, Study Chair — LeBonheur Children's Hospital
Locations (1):
- Le Bonheur Children's Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goulet O, Olieman J, Ksiazyk J, Spolidoro J, Tibboe D, Kohler H, Yagci RV, Falconer J, Grimble G, Beattie RM. Neonatal short bowel syndrome as a model of intestinal failure: physiological background for enteral feeding. Clin Nutr. 2013 Apr;32(2):162-71. doi: 10.1016/j.clnu.2012.09.007. Epub 2012 Sep 25. PMID 23159212
- [Background] Drenckpohl, D., et al., Adding Dietary Green Beans to Formula Resolves the Diarrhea Associated With a Bowel Resection in Neonates. ICAN: Infant, Child, & Adolescent Nutrition, 2013. 5(1): p. 8-13.
- [Background] Wessel J, Kotagal M, Helmrath MA. Management of Pediatric Intestinal Failure. Adv Pediatr. 2017 Aug;64(1):253-267. doi: 10.1016/j.yapd.2017.03.010. No abstract available. PMID 28688591
- [Background] Rabbani GH, Teka T, Zaman B, Majid N, Khatun M, Fuchs GJ. Clinical studies in persistent diarrhea: dietary management with green banana or pectin in Bangladeshi children. Gastroenterology. 2001 Sep;121(3):554-60. doi: 10.1053/gast.2001.27178. PMID 11522739
- [Background] Harvie ML, Norris MAT, Sevilla WMA. Soluble Fiber Use in Pediatric Short Bowel Syndrome: A Survey on Prevailing Practices. Nutr Clin Pract. 2018 Aug;33(4):539-544. doi: 10.1002/ncp.10089. Epub 2018 May 16. PMID 29767462
- [Background] Drenckpohl D, Hocker J, Shareef M, Vegunta R, Colgan C. Adding dietary green beans resolves the diarrhea associated with bowel surgery in neonates: a case study. Nutr Clin Pract. 2005 Dec;20(6):674-7. doi: 10.1177/0115426505020006674. PMID 16306306
- [Background] Homann HH, Kemen M, Fuessenich C, Senkal M, Zumtobel V. Reduction in diarrhea incidence by soluble fiber in patients receiving total or supplemental enteral nutrition. JPEN J Parenter Enteral Nutr. 1994 Nov-Dec;18(6):486-90. doi: 10.1177/0148607194018006486. PMID 7602722
- [Background] Becker B, Kuhn U, Hardewig-Budny B. Double-blind, randomized evaluation of clinical efficacy and tolerability of an apple pectin-chamomile extract in children with unspecific diarrhea. Arzneimittelforschung. 2006;56(6):387-93. doi: 10.1055/s-0031-1296739. PMID 16889120
- [Background] Koruda MJ, Rolandelli RH, Settle RG, Saul SH, Rombeau JL. Harry M. Vars award. The effect of a pectin-supplemented elemental diet on intestinal adaptation to massive small bowel resection. JPEN J Parenter Enteral Nutr. 1986 Jul-Aug;10(4):343-50. doi: 10.1177/0148607186010004343. PMID 3747092
- [Background] Rabbani GH, Teka T, Saha SK, Zaman B, Majid N, Khatun M, Wahed MA, Fuchs GJ. Green banana and pectin improve small intestinal permeability and reduce fluid loss in Bangladeshi children with persistent diarrhea. Dig Dis Sci. 2004 Mar;49(3):475-84. doi: 10.1023/b:ddas.0000020507.25910.cf. PMID 15139502
- [Background] Nakao M, Ogura Y, Satake S, Ito I, Iguchi A, Takagi K, Nabeshima T. Usefulness of soluble dietary fiber for the treatment of diarrhea during enteral nutrition in elderly patients. Nutrition. 2002 Jan;18(1):35-9. doi: 10.1016/s0899-9007(01)00715-8. PMID 11827762